CLINICAL TRIAL: NCT07313397
Title: Nurse-led and GP-supported Self-management Interventions to Reduce Cardiovascular Risks in Breast Cancer Survivors With Cardiovascular Diseases
Brief Title: Self-management Interventions to Reduce Cardiovascular Risks in Breast Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Queensland (Other)
Responsible Party: Principal Investigator, Anu Correya, Principal Investigator, University of Southern Queensland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ETH2025-0291
Record Dates: First submitted 2025-11-13; First posted 2025-12-31 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cardiovascular disease; Self-management Interventions; Breast Cancer Suvivors
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-management intervention group (Experimental): A combined face-to-face and telehealth self-management intervention will be conducted over four weeks, following assessment of the patients' cardiac condition, breast cancer, health literacy, and access to resources. The interventions will be carried out mainly by nurses, GPs, and allied health professionals, who will be included if needed. Patients and caregivers will be involved in the sessions. The self-management interventions will be behaviour change interventions, such as physical exercise, dietary modifications, smoking cessation and weight management.
  Interventions: Other: Self-management Interventions

INTERVENTIONS:
Other: Self-management Interventions — Self-management interventions will cover physical activity, smoking cessation, weight management, diet modifications, eliminate or reduce alcohol consumption and mind-body exercise such as taichi, yoga.

SUMMARY:
The goal of this proposed single-group pre-post pilot study is to assess the feasibility and acceptability of the codesigned Nurse-led and GP-supported self-management interventions (NGPS) to reduce cardiovascular risks in breast cancer survivors with cardiovascular diseases. The study will also assess the preliminary effects of the NGPS intervention on various outcomes, such as behavioural, physiological, psychological, and healthcare usage. These outcomes will be measured at three time points, which include the baseline measurement at recruitment (T1-week 1), right after the four weeks' intervention (T2-week 4), and eight weeks after completing the intervention (T3-week 12). The study will be conducted in the primary care centres, and the self-management interventions are behavioural change interventions such as physical activity, diet modifications, tobacco cessation, weight management, eliminating or reducing alcohol consumption, and mind-body exercises such as yoga. The main questions it aims to answer are:

1. What are the recruitment, retention, attrition, and completion rates of participants and potential adverse effects related to the NGPS interventions for the participants throughout the pilot study?
2. What are the adherence rates of the NGPS protocol, participants' response and completion rates of the study instruments during the data collection period of the pilot study?
3. Do this pilot study results indicate any significant differences in cardiovascular health outcomes (e.g., BMI and blood pressure), physical activity, dietary intake, QoL, self-efficacy, anxiety and depression between and across different time points (Baseline (T1), post-intervention (T2), follow-up (T3))?

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* confirmed diagnosis of breast cancer at stage I, II, or IIIa
* confirmed diagnosis of CVDs, including heart failure, coronary artery disease, stroke, or transient ischemic attack
* able to read, write, and communicate in English
* have completed active anticancer treatment including chemotherapy and radiotherapy, and are receiving regular healthcare in a primary care centre from GP/practice nurses and are willing to participate in the research study and provide informed consent.

Exclusion Criteria:

* patients with unstable health conditions with mental health issues or critically ill patients unable to participate in physical activities (e.g., suffering from life-threatening diseases, extremely weak), cognitive impairment, currently involved in another research study, or scheduled anticancer treatment during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer survivors
Enrollment: 15 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Baseline Information | Once at baseline
  Collect socio-demographic characteristics of the breast cancer survivors such as age, height, race/ethinicity, religion, education level, marital status, employment status and annual household income as well as medical history
Feasibility of recruitment | From recruitment start (Day 1 of the recruitment) to recruitment close (the day that the target sample reached), up to 12 months
  Number of weeks/months needed to reach target sample size
Recruitment rate | Recruitment rate will be assessed monthly over the recruitment period (up to 12 months).
  The percentage of eligible (or approached) participants who actually agree to take part in the study.
Retention rate | Across the entire trial period, from enrolment to eight weeks post study follow-up
  The percentage of participants who remain in the study
Dropout rate | Across the entire trial period, from enrolment to eight weeks post study follow-up
  The percentage of participants dropped out after the study enrolment
Feasibility of the questionnaires | Across the entire trial period, from enrolment to eight weeks post study follow-up
  The percentage of missing responses for each item and the entire scale in each questionnaires
Feasibility and acceptability of the study intervention- Adherence rate | From week one to week four, during the intervention period
  The percentage of participants who followed the prescribed interventions as intended
Safety of the intervention- Adverse Events related to the Nurse-led and GP-supported self-management (NGPS) intervention | From week one to week four, during the intervention period
  Asking the participants to record any discomfort feelings or adverse events related to the NGPS intervention, keeping daily logbook and report via telephone or face-to-face
Acceptability of the intervention | At eight-week follow up
  Feedback on the NGPS program will be gained by using an investigator-created questionnaire. Participants are asked to specify the extent to which they agree with each statement about the intervention by selecting one response option that best indicates their views. The numeric value will range from 1 to 5, where 1 indicates strongly disagree, 2 indicates disagree, 3 indicates neither agree nor disagree, 4 indicates agree, and 5 indicates strongly agree. The minimum value is 1, and the maximum score is 5. Higher scores indicate greater acceptability of the intervention and a better outcome.

SECONDARY OUTCOMES:
Physiological outcomes- BMI | At baseline (T1), immediately post intervention (T2), and eight-week follow-up (T3)
  Measuring weight in kilograms, height in centimeters and height and weight will be combined to report BMI in kg/m^2.
Physiological outcomes-blood pressure | At baseline (T1), immediately post intervention (T2), and eight-week follow-up (T3)
  Measuring blood pressure in millimeters of mercury.
Physiological outcomes-heart rate | At baseline (T1), immediately post intervention (T2), and eight-week follow-up (T3)
  Measuring heart rate in beats per minute.
Behavioural outcomes using 15-item food frequency questionnaire | At baseline (T1), immediately post intervention (T2), and eight-week follow-up (T3)
  Behavioural outcome-dietary outcome Dietary outcomes: dietary intake will be measured by using a 15-item Food Frequency Questionnaire. This food frequency questionnaire is widely used in cardiac patients to screen for poor dietary patterns and has an overall good agreement with the diet history. This has been tested in female patients. The dietary intake was captured using frequency-based units with participants reporting their usual consumption of key food groups. The participants will be asked to mark each component on the 15-item food frequency questionnaire to best reflect their dietary pattern based on the scoring system on the scale. During analysis, a summary diet quality score will be calculated, with higher scores indicating better outcomes and healthier dietary patterns.
Behavioural outcomes- Self-reported smoking status | At baseline (T1), immediately post intervention (T2), and eight-week follow-up (T3)
  Behavioural outcome- smoking status Self-reported smoking status. Participants will be asked to report their smoking status by selecting one option that best describes them. The numeric values will be 0, 1 and 2. O indicates never smoked (have never smoked cigarettes or tobacco products), 1 indicates former smoker (previously smoked but does not currently smoke), and 2 indicates current smoker (currently smoke cogarettes or tobacco products). The minimum value will be 0, and the maximum value will be 2. Higher scores indicate a poor outcome or greater current exposure to smoking.
Behavioural outcomes-Physical activity assessment using the International Physical Activity Questionnaire | At baseline (T1), immediately post intervention (T2), and eight-week follow-up (T3)
  Behavioural outcome-Physical activity Physical activity: it will be measured by using the International Physical Activity Questionnaire (IPAQ). This IPAQ is a well-validated tool in Australian adults and has good reliability and validity for assessing physical activity in breast cancer survivors. IPAQ data will be collected minutes per day or hours per day and converted to MET-minutes per week for analysis. Responses will be scored and classified according to established IPAQ scoring guidelines into one numeric value of 1-3 based on reported frequency, duration, and intensity of physical activity. The numeric value of 1 indicates low physical activity, 2 indicates moderate physical activity, and 3 indicates high physical activity. The minimum value is 1, and the maximum value is 3. Higher scores indicate better outcomes or greater levels of physical activity.
Psychological outcome-Self efficacy | At baseline (T1), immediately post intervention (T2), and eight-week follow-up (T3)
  Psychological outcome:
  Self-efficacy: It will be measured by using the General Self-Efficacy Scale (GSES). This 10-item scale will measure patients' beliefs in their ability to cope with various challenging situations. GSES demonstrated high reliability and validity across a range of populations. The GSES uses a 4-point Likert response scale yielding a total score ranging from 10 to 40, with higher score indicating greater self efficacy.
Psychological outcomes-Quality of Life | At baseline (T1), immediately post intervention (T2), and eight-week follow-up (T3)
  Psychological outcome:
  Quality of life (QoL): It will be measured by using the Functional Assessment of Cancer Therapy-Breast (FACT-B). This is a targeted QoL measurement tool for breast cancer patients with satisfactory reliability and validity. This tool will assess physical well-being, social well-being, emotional well-being and functional well-being, as well as 10 items for additional concerns. The FACT-B uses a 5-point Likert response scale (0-4)across its subscales, with the summed score representing breast cancer specific QoL.
Psychological outcome-Anxiety and Depression | At baseline (T1), immediately post intervention (T2), and eight-week follow-up (T3)
  Psychological outcome:
  Anxiety and depression: They will be measured by using the well-established 14-item Hospital Anxiety and Depression Scale (HADS). HADS is a widely adopted tool in various populations, including cancer patients and primary healthcare settings. The HADS uses a 4-point Likert scoring system (0-3), yielding subscale scores from 0-21 for anxiety and depression.
Healthcare usage | From week one to week four, during the intervention period and at eight week follow-up
  When a participant uses health services related to the cardiovascular conditions such as hospital visits and GP visits will be recorded using an investigator created logbook.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Wang, PhD, Principal Investigator — University of Southern Queensland
Locations (3):
- Australia (3):
  - Greens Medical Group, Dandenong South, Melbourne, Victoria
  - Keys Medical Centre, Keysborough, Melbourne, Victoria
  - TLC Medical Clinic, Noble Park, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No